CLINICAL TRIAL: NCT00002007
Title: A Pilot Trial Evaluating an Alternating Schedule of Recombinant Human GM-CSF and Azidothymidine in Patients With HIV Infection and Leukopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 067C; 202
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: HIV Infections; Cytopenias
Keywords: Leukopenia; Granulocyte-Macrophage Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Leukopenia; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; sargramostim

INTERVENTIONS:
Drug: Zidovudine
Drug: Sargramostim

SUMMARY:
To evaluate the safety of repeated courses of sargramostim ( recombinant granulocyte-macrophage colony-stimulating factor; GM-CSF ) administered subcutaneously to patients with HIV infection and leukopenia. To determine if administration of GM-CSF will prevent some or all of the hematologic toxicity associated with zidovudine ( AZT ) treatment in patients with pre-existing leukopenia. To assess any clinical and/or virologic benefits from administering alternating weeks of GM-CSF and AZT to patients with symptomatic HIV infection who have a history of cytologically confirmed Pneumocystis carinii pneumonia ( PCP ) or a circulating absolute CD4 lymphocyte count less than 200 cells/mm3.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serum antibody to HIV with or without evidence of HIV antigenemia.
* White blood cells (WBC) = or < 4500 cells/mm3 measured on at least 2 occasions separated by a minimum of 1 week.
* Qualifying indications for AZT therapy.
* Life expectancy = or > 6 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Current or past history of malignancy including Kaposi's sarcoma.
* Excessive diarrhea or significant malabsorption.
* If patients have had > 10 percent weight loss within the past 3 months, they should not have malabsorption as evidenced by serum carotene < 75 IU/ml, serum vitamin A < 75 IU/ml, significant malabsorption 4 foul-smelling or greasy stools per day or other criteria.
* Currently hospitalized or hospitalized within the last 4 weeks for the treatment of opportunistic infection (IO).
* Less than 1 week since completing treatment of Pneumocystis carinii pneumonia (PCP).
* Active OI requiring systemic treatment.
* Evidence of nutritional deficiencies that may contribute to anemia and/or leukopenia.

Concurrent Medication:

Excluded within 4 weeks of study entry:

* Zidovudine (AZT).
* Other antiviral agent associated with leukopenia.
* Investigational drug.
* Immunomodulators.
* Interferon.
* Steroids.
* Excluded within 8 weeks of study entry:
* Ribavirin.
* Excluded within 4 months of study entry:
* Suramin.

Patients with the following are excluded:

* Current or past history of malignancy including Kaposi's sarcoma.
* Excessive diarrhea or significant malabsorption.
* Currently hospitalized or hospitalized within the last 4 weeks for the treatment of opportunistic infection (OI).
* Less than 1 week since completing treatment of Pneumocystis carinii pneumonia (PCP).
* Evidence of nutritional deficiencies that may contribute to anemia and/or leukopenia.

Prior Medication:

Excluded:

* Prophylactic therapy for Pneumocystis carinii pneumonia (PCP) that may cause leukopenia.

Risk Behavior:

Excluded:

* Current drug or alcohol abusers.
* Unprotected sexual contact or other activities that may result in reinfection with HIV.

Patients must be willing to refrain from unprotected sexual contact or other activities that may result in reinfection with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Natl Cancer Institute, Bethesda, Maryland, United States